CLINICAL TRIAL: NCT05004818
Title: Galvanic Vestibular Stimulation as a Novel Treatment for Seasickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDF 1298-2013
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Motion Sickness; Seasickness; Habituation; Vestibular Time Constant
Keywords: Motion Sickness; Seasickness; Galvanic vestibular stimulation; Rotatory chair; Vestibular time constant
MeSH Terms: conditions — Motion Sickness; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham procedure (Sham Comparator): Participants with severe motion sickness were sited in the the rotatory chair with the videonystagmography recorder masking their eyes, while two galvanic vestibular stimulation electrodes were connected to the mastoid processes. No active stimulus was given.
  Interventions: Procedure: Sham procedure
- GVS stimulation coupled with inverse phase rotatory chair stimulation (Experimental): Participants with severe motion sickness were sited in the the rotatory chair with the videonystagmography recorder masking their eyes, while two galvanic vestibular stimulation electrodes were connected to the mastoid processes. The rotatory chair was activated in sinusoidal harmonic acceleration protocol in inverse phase to galvanic vestibular stimulation.
  Interventions: Procedure: GVS stimulation coupled with inverse phase rotatory chair stimulation at sinusoidal harmonic acceleration protocol

INTERVENTIONS:
Procedure: GVS stimulation coupled with inverse phase rotatory chair stimulation at sinusoidal harmonic acceleration protocol — GVS stimulation coupled with inverse phase rotatory chair stimulation at sinusoidal harmonic acceleration protocol
  Arms: GVS stimulation coupled with inverse phase rotatory chair stimulation
Procedure: Sham procedure — Participants with severe motion sickness were sited in the the rotatory chair with the videonystagmography recorder masking their eyes, while two galvanic vestibular stimulation electrodes were connected to the mastoid processes. No active stimulus was given.
  Arms: sham procedure

SUMMARY:
subjects with severe seasickness, who failed to habituate to sea conditions after at least six month of active sailing, were enrolled to the single-blind randomized control study. The intervention group was treated with rotatory chair stimulation at sinusoidal harmonic acceleration protocol coupled with galvanic vestibular stimulation to the mastoid processes. This unique procedure was hypothesized to promote habituation to seasickness. The control group underwent a sham procedure. All study participants filled out seasickness questionnaires at set time points following the intervention and underwent repeated step testing to determine their vestibular time constant. The number of anti-motion sickness clinic visits and scopolamine prescriptions was also recorded in the three months period following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* maximum score of 7 on the Wiker seasickness questionnaire in moderate sea conditions, with wave height of 0 - 1.5 m
* All had been sailing regularly for at least six months before enrolling in the study

Exclusion Criteria:

* history of hearing loss
* otoscopic findings of ear pathology
* an implanted electrode
* a finding of vestibulopathy on otoneurologic examination
* withdrawal by any subject of his informed consent.

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Vestibular time constant | Until one month following the intervention
  Vestibular time constant was measured using repeated rotatory chair stimulation in step protocol.
Seasickness severity | Until one month following the intervention
  Seasickness severity as determined by Wiker questionnaire at set time frames following the intervention
scopolamine drug prescription | Until three months following the intervention
  scopolamine drug prescriptions were calculated for each participant and compared between the two groups
Anti-motion sickness clinic visits | Until three months following the intervention
  Anti-motion sickness clinic visits were calculated for each participant and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Dror Tal, PhD, Principal Investigator — The Israel Naval Medical Institute, IDF Medical Corps, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutkovich YE, Lagami D, Jamison A, Fonar Y, Tal D. Galvanic vestibular stimulation as a novel treatment for seasickness. Exp Brain Res. 2022 Feb;240(2):429-437. doi: 10.1007/s00221-021-06263-w. Epub 2021 Nov 15. PMID 34782915